CLINICAL TRIAL: NCT01585571
Title: Observational Study of Balance and Posture in Adults With Cerebral Palsy
Brief Title: Balance and Posture in Adults With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: R01HD069769 (NIH)
Record Dates: First submitted 2012-04-18; First posted 2012-04-26 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
Keywords: Balance; Posture; Virtual Environment; Cerebral Palsy; Adults
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: 50 individuals of typical development with no known neuromuscular issues.
- Adults with CP: 50 Individuals with a pediatric diagnosis of spastic, hemiplegic, diplegic or quadriplegic cerebral palsy.

SUMMARY:
The results of this study will have an impact upon public heath policy as adults with cerebral palsy (CP) present a growing and underserved population in the United States. At the conclusion of this study, we will have identified the means by which the adult with CP maintains their upright position, which is essential for activities of daily living and for movement. With this knowledge, it will be possible to develop clinical and rehabilitation interventions that will improve their arm and leg function, and reduce the risk of falls for the adult with CP.

DETAILED DESCRIPTION:
Individuals with Cerebral Palsy (CP) present with considerable functional heterogeneity, and demonstrate a marked decrease in functional status with age due to the development of disturbances in somatosensory function, secondary neuromuscular impairments, and poor control over the trunk muscles. These factors promote balance instability, result in an increased fall risk, and contribute to lost functional capabilities. Little is known about the progression of neuromotor and somatosensory impairments as individuals with CP age, thus a knowledge gap exists concerning postural control and balance in the adult with CP, particularly which those associated with aging (primary) and those associated with compensatory behaviors. The objective of this proposal is to explore mechanisms behind abnormal motor response in postural control in the adult with CP. We HYPOTHESIZE that somatosensory reliance, as well as muscle passive and active properties, change with aging and functional adaptation. In order to address our central hypothesis, we propose the following specific aims: SPECIFIC Aim 1: To examine the central disturbances of sensory processing and sensorimotor integration that contribute to abnormal postural control in young adults with CP. We will: a) determine the effect of visual dependence on postural control in the adult with CP as directly measured with a test for visual dependence; and b)relate the presence of visual dependence to the effect of disturbances of the visual flow field on the center of mass (CoM) and center of pressure (CoP) responses in the adult with CP; and c) determine the relationship between central disturbances of sensory processing and sensorimotor integration on functional balance as measured by standardized clinical assessments of balance and fall risk. SPECIFIC Aim 2: To examine the peripheral alterations in passive muscle-tendon properties that could contribute to abnormal postural control in young adults with CP. We will determine the effects of a disturbance of the base of support, a disturbance to the visual flow field, and a combined disturbance of the two on joint kinematics,CoP, and CoM responses in the adult with CP using functional principal component (time-series) analyses. SPECIFIC Aim 3: To examine the impaired muscle activation and loss of selectivity over muscle control that contributes to abnormal postural control in young adults with CP. We will determine the effects of a disturbance of the base of support, a disturbance to the visual flow field, and a combined disturbance of the two on the surface electromyographic (sEMG) activity of lower limb and trunk muscles using wavelet analyses. At the conclusion of this study, we will have characterized postural control strategies employed by adults with CP in the presence of somatosensory and biomechanical perturbations. The combination of our innovative methodology to challenge all aspects of the sensorimotor system, with our analytical approach of both time series and wavelet analysis of the data, will allow us to separate the primary dynamic postural deficits from compensatory actions, a critical distinction for optimizing treatment interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with spastic diplegic or quadriplegic CP with the ability to stand for a period of 2 minutes
* Cognitive/communication skills sufficient to follow multiple step commands and to attend to tasks associated with data collection
* The control group will consist of age matched adults with no known neurological or somatosensory impairments.
* Subjects in all groups cannot have a reported sensitivity to motion sickness or visual field deficits or visual problems (lower than 20/40) not corrected by glasses.

Exclusion Criteria:

* Abnormal score for vestibular integrity as tested with the Dynamic Illegible 'E'-test
* Abnormal sensation to light touch and kinesthesia in the foot and ankle as assessed using the monofilament test.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The proposed investigation will be a cross-sectional study conducted with adolescents and young adults with typical development, and adolescents and young adults classified as having spastic diplegic or spastic quadriplegic CP between 15 and 30 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Center of Mass and Center of Pressure | 4 hours
  The investigators will measure the movement of the subject's center of mass and center of pressure using a force platform while they are looking at different visual scenes and with slow force plate movements.

SECONDARY OUTCOMES:
Muscle activity | 4 hours
  Muscle activity (recording using surface electrodes) will be performed while subjects are looking at different visual scenes and with slow force plate movements.
Movement of the legs and trunk | 4 hours
  Movement of the knee, ankle, hip and trunk (recorded using surface mounted markers) will be performed while subjects are looking at different visual scenes and with slow force plate movements.
Visual dependence | 1 hour
  Subjects will be seated in a chair, and asked to align a rotating rod to a vertical or horizontal position while receiving conflicting visual information ( a box placed around the rod in an off-center position)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lauer, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, VEPO Laboratory, Philadelphia, Pennsylvania, United States